CLINICAL TRIAL: NCT05675735
Title: Leveraging Regulatory Flexibility for Methadone Take-Home Dosing to Improve Retention in Treatment for Opioid Use Disorder: A Stepped-Wedge Randomized Trial to Facilitate Clinic Level Changes
Brief Title: Leveraging Regulatory Flexibility for Methadone Take-Home Dosing to Improve Retention in Treatment for Opioid Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-00892
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Problems Related to Social Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): 6 of the 36 recruited opioid treatment programs (OTPs) will be enrolled in group 1. Group 1 will start the six-month intervention at Baseline and end at Month 6.
  Interventions: Behavioral: Clinic-Level Multidimensional Intervention
- Cohort 2 (Experimental): 6 of the 36 recruited opioid treatment programs (OTPs) will be enrolled in Cohort 2. Cohort 2 will start the six-month intervention at Month 6 and end at Month 12.
  Interventions: Behavioral: Clinic-Level Multidimensional Intervention
- Cohort 3 (Experimental): 6 of the 36 recruited opioid treatment programs (OTPs) will be enrolled in Cohort 3. Cohort 3 will start the six-month intervention at Month 12 and end at Month 18.
  Interventions: Behavioral: Clinic-Level Multidimensional Intervention
- Cohort 4 (Experimental): 6 of the 36 recruited opioid treatment programs (OTPs) will be enrolled in Cohort 4. Cohort 4 will start the six-month intervention at Month 18 and end at Month 24.
  Interventions: Behavioral: Clinic-Level Multidimensional Intervention
- Cohort 5 (Experimental): 6 of the 36 recruited opioid treatment programs (OTPs) will be enrolled in Cohort 5. Cohort 5 will start the six-month intervention at Month 24 and end at Month 30.
  Interventions: Behavioral: Clinic-Level Multidimensional Intervention
- Cohort 6 (Experimental): 6 of the 36 recruited opioid treatment programs (OTPs) will be enrolled in Cohort 5. Cohort 5 will start the six-month intervention at Month 30 and end at Month 36.
  Interventions: Behavioral: Clinic-Level Multidimensional Intervention

INTERVENTIONS:
Behavioral: Clinic-Level Multidimensional Intervention — The proximal goal of the intervention will be to increase OTP uptake of flexible THD. The intervention addresses facilitators and barriers to THD practices as identified by existing studies as well as those found during the first phase of the current project. The intervention will be designed to address the information gaps, training needs, and beliefs of individuals across the organizations.

SUMMARY:
Using a stepped-wedge randomized controlled trial, the study will test whether a clinic-level multidimensional intervention conducted in 36 opioid treatment programs (OTPs) will improve clinical decision making, regulatory confusion, legal liability concerns, capacity for clinical practice change, and financial barriers to take- home dosing (THD) for methadone as compared to treatment as usual.

DETAILED DESCRIPTION:
Regulatory changes made during the COVID-19 public health emergency (PHE) that relaxed criteria for take- home dosing (THD) of methadone offer an opportunity to improve retention in care with a lifesaving treatment. Methadone is a highly effective medication for treating opioid use disorders (OUD) that is provided in opioid treatment programs (OTPs). Yet, longstanding regulatory restrictions limit the availability of methadone as well as create demands that heavily burden clients by requiring frequent visits to clinics. The rationale for these regulations is to safeguard against diversion and overdoses from methadone. Yet, the history and application of methadone regulations stem from stigmatized and racist notions of people with OUD. Most OTPs are located within communities with predominantly Black/African American or Latinx populations. Consequently, Black/African American and Latinx individuals have greater access to methadone than other, less restricted, medications for OUD. Within OTPs, Black/African American and Latinx individuals are less likely to receive adequate dosing levels of methadone and have lower retention than non-Hispanic White clients. More flexible THD may help address disparities in care. Currently, there is a national debate about balancing safety concerns over more flexible THD against the benefits of client retention and quality of life. Low offering of THD in many OTPs suggests a need for new data-driven interventions to encourage changes in engrained clinical workflows and long-standing stigmatizing beliefs about OUD clients. OTP leadership and staff express concern about misapplying regulatory flexibility, of iatrogenic effects of greater THD, and about legal liability from overdoses or diversion. Finally, financial concerns mount for organizations that have long based their business models on billing for frequent in-person medication dispensing. This project stems from a well-established academic-public partnership in New York State between the Office of Addiction Services and Supports (OASAS) and research collaborators from New York University, Cornell University, and the University of Connecticut. The investigators propose a two-part project to develop then test a multidimensional OTP intervention to address clinical decision making, regulatory confusion, legal liability concerns, capacity for clinical practice change, and financial barriers to THD. The intervention will include OTP THD specific dashboards drawn from multiple State databases. The approach will be informed by the Health Equity Implementation Framework. In year 1, the investigators will employ an explanatory sequential mixed method design to combine analysis of large state administrative databases-Medicaid, treatment registry, THD reporting-with qualitative interviews to refine the intervention. In years 2-5, the investigators will conduct a stepped-wedge trial with 36 OTPs (~10,800 Medicaid clients/yr) randomized to 6 cohorts of a six-month long clinic-level intervention over three years. The trial will test the effects of the intervention on 1) THD; 2) retention in care; and 3) adverse healthcare events. The investigators will specifically examine the effects of the intervention for Black/African American and Latinx clients.

ELIGIBILITY:
Inclusion Criteria:

* Clinic staff inclusion will include anyone who works at the 10 clinics that the OASAS client data system generates from the quantitative analysis in year one. In years 2-5, clinics chosen by the OASAS client data system will be placed into six cohorts. Only staff from these clinics will be eligible.
* Patient inclusion will include anyone aged 18 or older who has been receiving take-home methadone for at least 30 days.

Exclusion Criteria

• There are no exclusion criteria related to sex/gender to increase the generalizability of the findings. The investigators will note include children in this study because the treatment system that we are examining largely excludes adolescents and younger children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 7-Day THD Prescriptions | Pre-Intervention (from Baseline up to Month 30), Post-Intervention (from Month 6 up to Month 36)
  7-day THD is defined as a prescription to pick up doses of methadone every 7 days or less often.
Change from Baseline in 14-Day THD Prescriptions | Pre-Intervention (from Baseline up to Month 30), Post-Intervention (from Month 6 up to Month 36)
  14-day THD is defined as a prescription to pick up doses of methadone every 14 days or less often.
Change from Baseline in 28-Day THD Prescriptions | Pre-Intervention (from Baseline up to Month 30), Post-Intervention (from Month 6 up to Month 36)
  28-day THD is defined as a prescription to pick up doses of methadone every 28 days or less often.
Change from Baseline in OTP Care Retention | Pre-Intervention (from Baseline up to Month 30), Post-Intervention (from Month 6 up to Month 36)
  Will be calculated only among patients who have been in treatment for less than 12 months at the start of the study.
Change from Baseline in Number of Emergency Department Visits | Pre-Intervention (from Baseline up to Month 30), Post-Intervention (from Month 6 up to Month 36)
Change from Baseline in Number of Hospitalizations | Pre-Intervention (from Baseline up to Month 30), Post-Intervention (from Month 6 up to Month 36)
Change from Baseline in All-Cause Mortality | Pre-Intervention (from Baseline up to Month 30), Post-Intervention (from Month 6 up to Month 36)
  All-Cause Mortality defined as death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Neighbors, PhD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - University of Connecticut, Storrs, Connecticut
  - University at Buffalo, Buffalo, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Aggregate data will be reported to protect privacy of participants. Data will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Charles.Neighbors@nyulangone.The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposes to use the data will be granted access upon reasonable request. Requests should be directed to Charles.Neighbors@nyulangone. To gain access, data requestors will need to sign a data access agreement.